CLINICAL TRIAL: NCT06492278
Title: Open Pilot Trial of a Resiliency Group Program for Caregivers of Children With Learning and Attentional Difficulties: Supporting Parents Raising Kids (SPARK)
Brief Title: Resiliency Programming for Caregivers of Children With Learning and Attentional Difficulties
Acronym: SPARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Elyse Park, PhD, Professor of Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024P001219; 1R56AT011869-01A1 (NIH)
Record Dates: First submitted 2024-06-27; First posted 2024-07-09 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-01

CONDITIONS: Parenting; Stress; Learning Disabilities, Child; Attention Difficulties
Keywords: Resiliency training; Stress management; Learning and attentional disabilities
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SMART-3RP (Experimental): This is an adapted 8-session group program of the Relaxation Response Resiliency Program (3RP) for parents of children with LAD.
  Interventions: Behavioral: SMART-3RP
- Health Education Program (Active Comparator): This is an adapted 8-session group program to provide health behavior education.
  Interventions: Behavioral: Health Education Program

INTERVENTIONS:
Behavioral: SMART-3RP — The adapted program incorporates the three prongs of the 3RP: RR elicitation, stress awareness, and adaptive strategies.
  Arms: SMART-3RP
Behavioral: Health Education Program — This is a multiple behavior change program that addresses sleep, exercise, nutrition, substance use, and working with one's healthcare team.
  Arms: Health Education Program

SUMMARY:
This is a randomized open pilot trial enrolling up to 40 co-primary caregivers of children with LAD. Participants will be randomized to receive either mind-body resiliency group (SMART-LAD, intervention) or an evidence-based group intervention Health Education Program (HEP, control) which is a multiple behavior change program that addresses sleep, exercise, nutrition, substance use, and working with one's healthcare team. Both the SMART-3RP and HEP programs have been modified based on adaptions from our previous qualitative study.

DETAILED DESCRIPTION:
The primary objective of this protocol is to conduct an open pilot to elicit initial quantitative and qualitative feedback regarding feasibility and acceptability of the interventions (SMART-3RP and HEP) that we have refined. Both groups are designed to improve well-being for caregivers experiencing stress-related to caring for a child with LAD.

The investigators will ask participants to complete approximately 15-minute survey batteries via REDCap at baseline and after the 8-week program, including assessments of intervention feasibility and acceptability as well as psychosocial outcomes. To inform plans for ongoing program refinement, the investigators will also elicit specific feedback regarding study assessment tools, recruitment procedures, and group composition.

Results will be used to inform a larger randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Age 18 or older
* Ability to participate in group, virtual sessions including access to computer, tablet, or smartphone, and internet
* Parents or guardians of a child (< age 18) with LAD.

Exclusion Criteria:

* Parents with significant psychiatric conditions (i.e., active suicidality or psychosis) or who are otherwise unable to participate, at the investigators' clinical discretion.
* Only one parent per family can participate.
* Unwilling or unable to participate in the study
* Considered medically or otherwise unable to participate by the study PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Feasibility of the refined interventions (SMART-3RP and HEP) | Approximately 3 months (approximately 8-10 weeks after intervention start)
  Rates of intervention attendance (# of sessions), rates of participant recruitment (%) enrollment, survey completion rates (%).
Acceptability of the refined interventions (SMART-3RP and HEP) | Approximately 3 months (approximately 8-10 weeks after intervention start)
  Likert ratings of group comfort and cohesiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Elyse R Park, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No